CLINICAL TRIAL: NCT00178269
Title: A Phase Ii Clinical Study Using Weekly Low-Dose Taxotere® (Docetaxel) With Concurrent Radiotherapy For Localized, Inoperable Carcinoma Of The Uterine Cervix
Brief Title: Low-Dose Taxotere® (Docetaxel) With Concurrent Radiotherapy For Localized, Inoperable Carcinoma Of The Uterine Cervix
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Yuhchyau Chen, MD,Ph.D, University of Rochester. Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URCC 1328
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Cervix Neoplasm
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Docetaxel; Radiotherapy

INTERVENTIONS:
Drug: docetaxel
Procedure: Radiation Therapy

SUMMARY:
The purpose of this study is to find out how effectively cervix cancer is controlled when radiation is combined with low-dose chemotherapy (Taxotere) . The use of low-dose Taxotere, once per week, with radiation is a new treatment for cervical cancer. This study will also see how well this treatment regimen can be tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of squamous, adenocarcinoma, or adenosquamous carcinoma of the uterine cervix including FIGO (International Federation of Gynecologists and Obstetricians) stage IB to IVA with or without pelvic adenopathy.
* No evidence of para-aortic or distant metastases. Must have evaluable disease.
* Zubrod Performance Status 0-2 or Karnofsky Performance Status > 60
* Laboratory values must be as follows:

White blood cell count: > 3,000/mm3,Absolute granulocyte count: > 1,500/mm3, Hemoglobin > 8.0 g/dl, Platelets: > 100,000/mm3, Serum creatinine: < 2.5 mg/dl, Serum calcium: < 1.3 x institutional upper normal limit,Hepatic criteria as follows: Total Bilirubin < ULN for the institution,

* Signed study-specific informed consent p
* Age > 18 years.
* Peripheral neuropathy must be < grade 1.

Exclusion Criteria:

* Prior or simultaneous malignancies (other than skin cancer) unless disease-free
* Medical illness preventing the use of taxane-based chemotherapy.
* Carcinoma of the cervix with the following histology: melanoma, sarcoma, small carcinoid, glassy cell, clear cell, and adenoid cystic.
* Previous or current medical or psychiatric illness that would prevent informed consent
* Patients known to be infected with HIV or a history of AIDS are excluded.
* Prior surgery for carcinoma of the cervix other than a biopsy.
* Patients with para-aortic disease.
* Previous pelvic radiation therapy or systemic chemotherapy is not permitted.
* Women who are pregnant or breast-feeding are excluded from this study.
* Previous history of hypersensitivity reaction to Taxotere or other drugs formulated with polysorbate 80 must be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Primary Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuhchyau Chen, MD, Ph.D, Principal Investigator — Universtiy of Rochester, Dept of Radiation Oncology
Locations (1):
- University of Rochester, Dept. Radiation Oncology, Rochester, New York, United States